CLINICAL TRIAL: NCT01242306
Title: Head-to-Head Comparison of Endothelial Dysfunction (Bare Metal Stent vs Sirolimus Eluting Stent) in the Same Patient With Multiple Coronary Artery Lesions
Brief Title: Comparison of Endothelial Dysfunction (BMS vs SES) in the Same Patient With Multiple Coronary Artery Lesions
Acronym: CREDENTIAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Mischie Nicolae Alexandru, European Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREDENTIAL
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2009-04

CONDITIONS: Endothelial Dysfunction
Keywords: endothelial dysfunction acetylcholine bms ses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMS arm (Placebo Comparator): bare metal stent arm
  Interventions: Drug: intracoronary infusion of acetylcholine
- SES arm (Active Comparator): sirolimus eluting stent arm
  Interventions: Drug: intracoronary infusion of acetylcholine

INTERVENTIONS:
Drug: intracoronary infusion of acetylcholine — Acetylcholine will be infused at a concentration of 140 microg/minute, over a period of 2 minutes, yielding estimated intracoronary concentrations of 10(-5)mol/L, with the assumption of a flow rate of 80mL/min). All infusions will be delivered at a constant rate using an infusion pump. Subsequently, in order to evaluate the endothelium-independent vasomotor response, 2mg of isosorbide dinitrate or bolus 250microg of nitroglycerine will be infused by intracoronary bolus in all subjects. The response to nitrate will be recorded 1 minute after the bolus. A 3-min period will be allowed to elapse between each drug infusion.
  Other Names: cypher coroflex

SUMMARY:
This is a prospective, randomised study to compare the endothelial dysfunction of BMS vs SES, both implanted in the same patient with multiple de novo coronary artery lesions undergoing elective PCI. The primary end point will be the evaluation of endothelial dysfunction at 6 months follow-up by measuring the change in vessel diameter in 5 points of the stent and peri-stent site after infusion of acetylcholine.

DETAILED DESCRIPTION:
This prospective, randomised study compares the endothelial dysfunction of BMS vs SES, both implanted in the same patient with multiple de novo coronary artery lesions undergoing elective PCI. From february 2009 to may 2009 we aim to enroll 20 patients with at least two de novo significant angiographic stenoses in different coronary segments who will have similar diameter and length. The primary end point will be the evaluation of endothelial dysfunction at 6 months follow-up by measuring the change in vessel diameter in 5 points of the stent and peri-stent site after infusion of acetylcholine.

ELIGIBILITY:
Inclusion Criteria:

* stable angina pectoris
* at least two significant angiographic stenoses in different native coronary vessels or in the same vessel but two different ramifications with similar diameter
* non-surgical patients

Exclusion Criteria:

* acute coronary syndromes
* myocardial infarction within 3 months from event
* clinical or angiographic coronary vasospasm
* coronary angiographic findings of a fresh thrombus in the initial angiography (filling defect proximal to or involving the stenosis)
* coronary anatomy unsuitable for for intracoronary acetylcholine testing (left main coronary artery disease >30%, surgical three vessel disease or other anatomical considerations that make it unsafe to perform intracoronary studies)
* progression of lesions or development of de novo lesions in nontarget lesions or vessels on follow-up angiography
* patients with a vessel diameter < 2,50 mm and length lesions <10 and >30 mm.
* patients with vessel diameter difference (SES vs BMS) >0,5mm and length difference of the stenosis >50%
* lesions treated with balloon injury <10 mm or >50 mm in length
* severe left ventricular (LV) systolic dysfunction
* bifurcation/ostial
* presence of an unhealed dissection identified by intravascular ultrasound (IVUS) performed at the end of the study.
* angiographic restenosis in follow-up angiography
* patients with severe risk factors for endothelial dysfunction: severe renal failure, life expectancy less than 1 year, uncontrolled diabetes, uncontrolled hypertension (systolic blood pressure >180mmHg), currently smoking, uncontrolled hypercholesterolemia (total cholesterol >240mg/dl)
* any contraindication/nontolerance to the use of aspirin, heparin and/or clopidogrel
* lack of consent to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
evaluation of endothelial dysfunction at 6 months follow-up by measuring the change in vessel diameter in 5 points of the stent and peri-stent site after infusion of acetylcholine | 6 months
  evaluation of change in vessel diameters (vasoconstriction or vasodilatation) in proximal and distal stent territories, after intracoronary acetylcholine infusion, having as reference the baseline diameters, for the BMS artery vs the SES artery

CONTACTS AND LOCATIONS:
Overall Officials: Violini Roberto, MD, Study Chair — Azienda Ospedaliera San Camillo Forlanini; Mischie Nicolae Alexandru, MD, Principal Investigator — European Society of Cardiology; Nazzaro Marco, MD, Study Director — Azienda Ospedaliera San Camillo Forlanini
Locations (1):
- Azienda Ospedaliera San Camillo Forlanini, Roma, Roma, Italy

REFERENCES:
- [Derived] Mischie AN, Nazzaro MS, Fiorilli R, De Felice F, Musto C, Confessore P, Parma A, Boschetti C, Violini R. Head-to-head comparison of sirolimus-eluting stent versus bare metal stent evaluation of the coronary endothelial dysfunction in the same patient presenting with multiple coronary artery lesions: the CREDENTIAL study. Catheter Cardiovasc Interv. 2013 Sep 1;82(3):E184-91. doi: 10.1002/ccd.24844. Epub 2013 Mar 5. PMID 23359371